CLINICAL TRIAL: NCT01486368
Title: A Phase II Study of PF-03446962 in Patients With Advanced Malignant Pleural Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I207
Record Dates: First submitted 2011-12-01; First posted 2011-12-06 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Malignant Pleural Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — ascrinvacumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PF-03446962 (Experimental)
  Interventions: Drug: PF-03446962

INTERVENTIONS:
Drug: PF-03446962 — PF-03446962 will be administered by IV infusion every 2 weeks (q2w). A cycle will be 2 weeks in duration and include one administration of PF-03446962.

SUMMARY:
This is a non-randomized open label multicentre Phase II trial to evaluate the response rate of PF03446962 in patients with advanced malignant pleural mesothelioma who have been previously treated with cytotoxic chemotherapy.

DETAILED DESCRIPTION:
To assess the efficacy (response rate, complete and partial) of PF-03446962 given by IV infusion Day 1 of a 2 week cycle (14 days = 1 cycle) in patients with advanced malignant pleural mesothelioma and previously treated with cytotoxic therapy.

To assess the toxicity, safety and tolerability of PF-03446962.

To assess the duration of response or stable disease, stable disease rate, progression-free, median and overall survival rates.

To collect tissue and blood for banking and correlative science evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed malignant pleural mesothelioma.
* Patients must have advanced and/or metastatic disease, incurable by standard therapies.
* All patients must have a tumour block from their primary or metastatic tumour available and consent to release the block for correlative analyses. Centre/pathologist must have agreed to the submission of the specimens in both Stage I and II of accrual. For patients entered in Stage I of accrual, if no archival tissue is available, patient must undergo a biopsy prior to registration.
* All patients entered in Stage II of accrual must have an accessible tumour lesion (from primary or metastatic disease) for a fresh biopsy, which is formalin fixed and paraffin embedded. These patients must consent to this biopsy for entry on the trial.
* Presence of clinically and/or radiologically documented disease. At least one site of disease must be unidimensionally measurable as follows:
* Chest X-ray ≥ 20 mm CT scan (with slice thickness of ≤ 5 mm) ≥ 10 mm longest diameter Physical exam (using calipers) ≥ 10 mm Lymph nodes by CT scan ≥ 15 mm measured in short axis All radiology studies must be performed within 21 days prior to registration (Exception: Within 28 days if negative).
* Age ≥ 18 years.
* Patients must have a life expectancy of at least 12 weeks.
* ECOG performance status 0 or 1. Performance Status 2 patients are eligible, if, in the opinion of the investigator, they are suitable for inclusion in the study and are likely to be compliant with the study procedures (in particular the recommendations for supportive care and dose modification).

Previous Therapy

Cytotoxic Chemotherapy:

* Patients are eligible after first line cytotoxic chemotherapy has failed
* Patients must have received one, but no more than one, combination chemotherapy regimen for advanced disease, which must have contained a platinum agent, and treatment failure must have been documented

  o Exchange of one chemotherapy agent for another within a combination chemotherapy regimen due to toxicity (and not due to progressive disease) is not considered a new regimen in the following circumstances
  * Carboplatin is substituted for cisplatin due to nephrotoxicity or ototoxicity
  * One agent in the combination regimen is changed due to hypersensitivity occurring in the first cycle
* 28 days must have elapsed since last chemotherapy treatment (at least 6 weeks for nitrosoureas or mitomycin C) and patient must have recovered from toxic effects.

Other Anti-Cancer Therapy:

• Patients may have received other non-cytotoxic investigational therapy; 28 days must have elapsed since last treatment, such as anti-angiogenic or growth factor antagonists.

Radiation:

Patients may have had prior radiation therapy. A minimum of 28 days must have elapsed between the end of radiotherapy and registration onto the study. Radiation must have involved < 30% of functioning bone marrow and there must be measurable disease outside the previously irradiated area (patients whose sole site of disease is in previously irradiated area are ineligible) unless there is evidence of progression or new lesions have been documented, in the irradiated field). [Exceptions may be made however for low dose palliative radiotherapy].

Previous Surgery:

Previous major surgery is permitted provided that it has been at least 28 days prior to patient registration and that wound healing has occurred.

Laboratory requirements must be done within 7 days prior to registration) Hematology: Granulocytes (ANC) ≥1.5 x 109/L Platelets ≥100 x 109/L Chemistry: Bilirubin ≤ULN AST and ALT ≤2.5 x ULN Calcium ≤3 mmol /L INR ≤1.5 x ULN Serum creatinine ≤ULN Or Creatinine clearance ≥60 ml/min if creatinine is >ULN Creatinine clearance to be measured directly by 24 hour urine sampling or as calculated by Cockcroft Formula:Females: GFR=1.04 x(140-age)x weight in kg serum creatinine in μmol/L; Males: GFR=1.23 x (140-age)x weight in kg serum creatinine in μmol/L

* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to registration in the trial to document their willingness to participate.
* Patients must be accessible for treatment, response assessment and follow-up. Patients registered on this trial must be treated and followed at the participating centre. This implies there must be reasonable geographical limits (for example: 1 ½ hour's driving distance) placed on patients being considered for this trial. Investigators must assure themselves the patients registered on this trial will be available for complete documentation of the treatment, response assessment, adverse events and follow up.
* In accordance with NCIC CTG policy, protocol treatment is to begin within 2 working days of patient registration.

Exclusion Criteria:

* Patients with a history of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≥5 years.
* Patients with known brain metastases. (A head CT is not necessary to rule out brain metastases, unless there is clinical suspicion of CNS involvement). Patients with known brain metastases will be excluded from this trial due to their poor prognosis and their likelihood of developing progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to PF-03446962.
* Patients receiving concurrent treatment with other anti-cancer therapy or other investigational anticancer agents.
* Patients with any of the following cardiovascular findings are to be excluded:

  * QTc prolongation ( defined as a mean QTc interval with Bazetts correction equal to or greater than 470 msec) in screening ECG or history of familial long QT syndrome. An ECG must be done within 14 days prior to registration.
  * Patients with resting BP consistently higher than, systolic > 150 mmHg and/or diastolic > 100 mmHg (in the presence or absence of a stable dose of anti-hypertensive medication) or poorly controlled hypertension, history of labile hypertension or poor compliance with anti-hypertensive medication.
  * Patients who have experienced untreated and/or uncontrolled cardiovascular conditions and/or have symptomatic cardiac dysfunction (unstable angina, congestive heart failure, myocardial infarction within the previous year or cardiac ventricular arrhythmias requiring medication, history of 2nd or 3rd degree atrioventricular conduction defects). Patients with a significant cardiac history even if controlled, should have a LVEF > 50%.
* History of pulmonary embolism within the past 12 months; exceptions may be made for incidental pulmonary emboli found on routine scanning providing not within the past 6 months.
* History of cerebrovascular accident (CVA) or transient ischemic attack within 12 months prior to study entry.
* Patients with overt bleeding from any site (> 30 ml bleeding/episode) within 3 months of study entry are not eligible. No clinically relevant hemoptysis (> 5 ml fresh blood) within 4 weeks prior to study entry is permitted. Patients with only flecks of blood in sputum are permitted.
* Patients who require use of therapeutic doses of anticoagulants such as warfarin, heparin or low molecular weight heparin (except for low doses for prophylaxis). INR must be done within 7 days prior to registration.
* Patients with bowel obstruction or any condition or gastrointestinal tract disease that would increase the risk for gastrointestinal perforation, including abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days of treatment.
* Patients with serious illness or medical condition which would not permit the patient to be managed according to the protocol including, but not limited to:

  * History of significant neurologic or psychiatric disorder which would impair the ability to obtain consent or limit compliance with study requirements;
  * Active uncontrolled infection;
  * Any other medical conditions that might be aggravated by treatment;
  * Serious or non-healing wound, ulcer, or bone fracture.
* The following are exclusions for enrollment on the study:

  * Pregnant or lactating women. (N.B.: All women of childbearing potential must have a negative pregnancy test within 7 days prior to registration).
  * Women must be post-menopausal, surgically sterile or use two reliable forms of contraception while on study and for 6 months after discontinuing therapy. Men must be surgically sterile or use a barrier method of contraception with spermicide. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-06-26 (Actual); Primary Completion 2014-04-27 (Actual); Study Completion 2015-02-13 (Actual)

PRIMARY OUTCOMES:
Response Rate | 30 months
  Assessing the efficacy (response rate, complete and partial) of PF-03446962 given by IV infusion Day 1 of a 2 week cycle(14 days = 1 cycle) in patients with malignant pleural mesothelioma and previously treated with cytotoxic therapy.

SECONDARY OUTCOMES:
Amount and severity of adverse events | 30 months
  To assess toxicity, safety and tolerability of PF-03446962.
Duration of Response | 30 months
  To assess the duration of response or stable disease, stable disease rate, progression-free survival, median and overall survival rates
Blood and tissue marker evaluation | 30 months
  Specimen collection to look for markers in cancer cells. These markers might help predict which patients are most likely to be helped by the study drug PF-03446962.

CONTACTS AND LOCATIONS:
Overall Officials: Quincy Chu, Study Chair — Cross Cancer Institute, Edmonton, AB Canada; Paul Wheatley-Price, Study Chair — Ottawa Health Research Institute - General Division, Ottawa ON Canada
Locations (7):
- Canada (7):
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Ottawa Health Research Institute - General Division, Ottawa, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wheatley-Price P, Chu Q, Bonomi M, Seely J, Gupta A, Goss G, Hilton J, Feld R, Lee CW, Goffin JR, Maksymiuk A, Murray N, Hagerman L, Bradbury PA. A Phase II Study of PF-03446962 in Patients with Advanced Malignant Pleural Mesothelioma. CCTG Trial IND.207. J Thorac Oncol. 2016 Nov;11(11):2018-2021. doi: 10.1016/j.jtho.2016.06.024. Epub 2016 Jul 20. PMID 27449804